CLINICAL TRIAL: NCT04155125
Title: Open-Label Randomised Controlled Trial of Efepoetin Alfa for Treatment of Anaemia Associated With Chronic Kidney Disease Patients Not on Dialysis (ND-CKD). A Non- Inferiority Trial Compared to Methoxy Polyethylene Glycol-Epoetin Beta (MIRCERA)
Brief Title: A Study of Efepoetin Alfa in Treating Anaemia Associated With Chronic Kidney Diseases Patient
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PT Kalbe Genexine Biologics (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GXE4KGBio-001
Record Dates: First submitted 2019-10-29; First posted 2019-11-07 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Anaemia Associated With Chronic Kidney Disease
MeSH Terms: interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- efepoetin alfa (Experimental): Route of administration: Subcutaneous Injection.
  The administration interval and initial dosage for subjects who are randomly assigned to subcutaneous efepoetin alfa will be starting from 4 μg/kg BW once per 2 weeks, then titrated based on Hb level during study period.
  Interventions: Drug: efepoetin alfa
- Mircera (Placebo Comparator): Route of administration: Subcutaneous Injection.
  The starting dosage of Mircera arm will be 0.6 μg/kg BW per 2 weeks based on prior data in similar study populations with subsequent titration to achieve targeted Hb range. During the correction treatment period, the dosage of study drug will be adjusted to achieve a Hb level range within 10 - 12 g/dL and an increase ≥1.0 g/dL versus the individual patient's baseline Hb level. During the extension period, Hb levels should be maintained between 10 and 12 g/dL.
  Interventions: Drug: Mircera

INTERVENTIONS:
Drug: efepoetin alfa — The administration interval and initial dosage for subjects who are randomly assigned to subcutaneous efepoetin alfa will be starting from 4 μg/kg BW once per 2 weeks, then titrated based on Hb level during study period.
  Arms: efepoetin alfa
Drug: Mircera — The starting dosage of Mircera arm will be 0.6 μg/kg BW per 2 weeks based on prior data in similar study populations with subsequent titration to achieve targeted Hb range. During the correction treatment period, the dosage of study drug will be adjusted to achieve a Hb level range within 10 - 12 g/dL and an increase ≥1.0 g/dL versus the individual patient's baseline Hb level. During the extension period, Hb levels should be maintained between 10 and 12 g/dL.
  Arms: Mircera

SUMMARY:
This is an open-label, randomised, multicenter, Mircera-controlled, parallel-group, Phase III study to determine whether subcutaneous administered efepoetin alfa is as effective and well tolerated as subcutaneous Mircera for anaemia correction and maintenance in erythropoiesis stimulating agent (ESA)-naïve subjects who have CKD and are not on dialysis. ESA prior users who have stopped using ESA at least 12 weeks till screening will also be eligible for this study provided they fulfil all the subject entry criteria.

DETAILED DESCRIPTION:
The study will consist of a 20-week correction period for dosage titration and Hb correction, followed by an 8-week evaluation period for efficacy assessments of corrective treatment. Subjects who respond to efepoetin alfa (defined as an increase in Hb ≥1.0 g/dL versus baseline and Hb level within 10 - 12 g/dL range without blood transfusion during the 28 weeks after the first dose) will be eligible to continue treatment, and will be randomised to receive subcutaneous efepoetin alfa either once every 2W or every 4W for an additional 24-week extension period to assess long-term safety and maintenance effect. Mircera responders will also be allowed to continue the drug during the extension period, receiving it every 4 weeks using the dose equal to twice the previous once-every-two-week dose. The safety data collected will be part of an ongoing pooled analysis of safety data from the efepoetin alfa clinical development program.

ELIGIBILITY:
Inclusion Criteria:

1. Age should be greater than or equal to the minimum age of consent in the applicable country
2. Stage 3 or 4 CKD (eGFR ≥ 15 and < 60 mL/min/1.73 m2)
3. ESA-naive (no prior ESA use) subjects whose Hb at baseline is ≥ 8 g/dL and < 10 g/dL, or ESA prior users whose Hb at baseline is ≥ 8 g/dL and < 10 g/dL and who have stopped using ESA at least 12 weeks till the screening
4. Ferritin ≥ 100 ng/mL and transferrin saturation (TSAT) ≥ 20%
5. Subject must be willing to complete all study-related activities and follow-up visits
6. Evidence of a signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

1. Need for dialysis therapy expected in the next 12 months or rapid progression of CKD (e.g., eGFR decrease of >20% within 12 weeks)
2. Received a blood transfusion (including RBC transfusion) within the 12 weeks prior to screening, or blood transfusion is anticipated during the study period
3. Have a history of overt gastrointestinal bleeding or any other bleeding episode associated with a fall in Hb of ≥ 1 g/dL, within the last 8 weeks prior to screening
4. Have an unstable Hb for any reason, in the investigator's opinion
5. Have non-renal anaemia (any anaemia where the investigator considers the anaemia is predominantly due to a non-renal cause. Non-renal causes include, but are not limited to vitamin B12 or folic acid deficiency, homozygous sickle-cell disease, thalassemia of all types, other non-renal cause of anaemia such as myelodysplasia or haematological malignancies)
6. Platelet count of ≤ 50 x109/L
7. Vitamin B12 deficiency defined as total serum levels of < 181 pmol/L (246 pg/ml) 10
8. Folic acid deficiency defined as total serum levels < 7.63 nmol/L (3.37 ng/mL) 10
9. Pure red cell aplasia, or a history of pure red cell aplasia
10. Poorly controlled hypertension defined as a sitting SBP ≥170 mmHg and/or DBP ≥100 mm Hg
11. Chronic congestive heart failure (New York Heart Association class IV) or are otherwise at high risk for early withdrawal or interruption of the study (due to myocardial infarction, severe or unstable coronary artery disease, stroke, or severe liver disease) within the 12 weeks before screening or during screening
12. Active or not active malignancy (except non-melanoma skin cancer) within five years before screening
13. Planned live kidney transplantation scheduled within 52 weeks after the screening visit
14. Uncontrolled hyperparathyroidism, in the investigator's opinion
15. Uncontrolled hypothyroidism determined by the investigator that they cannot participate in the study
16. Active acute or chronic infection, or uncontrolled or symptomatic inflammatory disease (e.g., rheumatoid arthritis, systemic lupus erythematosus), or a C-reactive protein level > 15 mg/L. (Routinely screening for hepatitis B virus (HBV), hepatitis C virus (HCV), and human immunodeficiency virus (HIV) infection is not required in this protocol. By history or current clinical evidence, patients with active acute HBV or HCV infection should be excluded. Chronic HBV/HCV infection with LFTs > 3 times of normal are excluded. Known HIV positive patients are excluded)
17. Immunosuppressive therapy (other than corticosteroids for a chronic condition, or tacrolimus/cyclosporine) within 12 weeks prior to baseline
18. Life expectancy of less than 52 weeks
19. Planned surgery during the study period (excluding minor skin excisions)
20. Have received investigational drug(s) other than those of this study within 4 weeks prior to screening, or will receive investigational drug(s) other than those of this study during the study period
21. History or clinical evidence of cardiovascular, haematologic or hepatic (ALT, AST, bilirubin values above three times the upper limit of normal [ULN] at screening) or any physical conditions that, in the opinion of the investigator, would compromise participation in the study
22. With a cognitive or psychiatric condition rendering the subject unable to be cooperative with and complete study requirements
23. Hypersensitivity to any one of the investigational drugs
24. Subjects are, in the judgement of the investigator, otherwise inappropriate for entry into the study
25. Subjects who are investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the Investigator, or subjects who are KGBio or CRO employees directly involved in the conduct of the trial
26. Participation in other studies involving same investigational drug(s) (Phases 1-4) of this study within 12 weeks before screening
27. Females of childbearing potential or males who are unable/unwilling to take adequate contraceptive precautions defined by the protocol for the duration of the study and for at least 28 days after last dose of investigational product. Females have a positive pregnancy test result within 24 hours prior to study entry, is otherwise known to be pregnant, plans to become pregnant in the next 12 months or is currently breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of efepoetin alfa in the treatment of anaemia associated with CKD as measured by haemoglobin (Hb) response rate at the end of correction treatment evaluation period | Measurement from the date of Randomization till the End of the Corrective Treatment period, assessed up to 20 weeks.
  Measurement is done by an increase in Hb more than or equal to 1 g/dL compared with baseline and a Hb concentration within range of 10 - 12 g/dL inclusive without transfusion during evaluation period

SECONDARY OUTCOMES:
Characterise safety and tolerability of subcutaneous efepoetin alfa is being measured by based on the frequency of adverse events and on the number of out of range laboratory values. | Measurement from the time the subject provides informed consent through and including 28 calendar days after the last study drug administration.
  Safety endpoints parameters including Serious Adverse Events (SAE) specified below
  1. Composite outcome of cardiovascular death or a nonfatal myocardial infarction or stroke
  2. All-cause mortality
  3. Cardiovascular mortality
  4. Acute myocardial infarction
  5. Heart failure
  6. Acute kidney injury defined according to Acute Kidney Injury Network (AKIN) criteria
  7. Abnormal clinical laboratory tests (haematology, biochemistry including serum ferritin and TSAT)
  8. Anti-efepoetin alfa or anti-Mircera antibody titres
  9. Clinically meaningful abnormal findings of vital signs
  10. Development of clinically meaningful electrocardiogram abnormalities
  11. Hospitalisations (excluding those for logistic reasons)
  It is a composite outcome. Any abnormal test findings during the study will be helpful in reviewing the outcome.

CONTACTS AND LOCATIONS:
Locations (55):
- Australia (3):
  - Renal Research Gosford, Gosford, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Launceston General Hospital, Launceston, Tasmania
- Indonesia (6):
  - Rspad Gatot Soebroto, Jakarta Pusat
  - Rumah Sakit Islam Jakarta Cempaka Putih, Jakarta Pusat
  - Rumah Sakit Islam Jakarta Pondok Kopi, Jakarta Pusat
  - Rumah Sakit Pgi Cikini, Jakarta Pusat
  - Rumah Sakit Umum Pusat Fatmawati, Jakarta Pusat
  - Rumah Sakit Umum Pusat Nasional Dr Cipto Mangunkusumo, Jakarta Pusat
- Malaysia (9):
  - Seri Manjung Hospital, Seri Manjung, Perak
  - University of Malaya Medical Centre, Kuala Lumpur, Selangor
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Kajang, Kajang
  - Hospital Raja Perempuan Zainab II, Kota Bharu
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Hospital Serdang, Serdang
  - Hospital Sibu, Sibu
- Philippines (7):
  - M3 Dialysis Center, Bacolod City
  - Baguio General Hospital Medical Center, Baguio City
  - Norzel Medical and Diagnostic Clinic, Cebu City
  - De La Salle Medical and Health Sciences Institute, Dasmariñas
  - Davao Doctors Hospital, Davao City
  - West Visayas State University Hospital, Iloilo City
  - National Kidney and Transplant Institute, Quezon
- South Korea (9):
  - Chungnam National University Hospital, Daejeon
  - Korea University Ansan Hospital, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - The Catholic University of Korea Incheon St. Mary'S Hospital, Incheon
  - Chungnam National University Sejong Hospital, Sejong
  - Kyung Hee University Hospital At Gangdong, Seoul
  - The Catholic University of Korea Eunpyeong St. Mary'S Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary'S Hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary'S Hospital, Seoul
- Taiwan (15):
  - Changhua Christian Hospital, Changhua
  - Hualien Tzu Chi Hospital, Hualien City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Hospital, Kaohsiung City
  - Keelung Chang Gung Memorial Hospital, Keelung
  - Taiching Veterans General Hospital, Taichung
  - Kuang Tien General Hospital, Taichung
  - Chi Mei Medical Center, Tainan
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Far Eastern Memorial Hospital, Taipei
  - Taipei Medical University - Shuang Ho Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Thailand (6):
  - Vajira Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Thammasat University Hospital, Pathum Thani
  - Songklanagarind Hospital, Songkhla
  - Sunpasitthiprasong Hospital, Ubon Ratchathani